CLINICAL TRIAL: NCT05448937
Title: Clinical And Radiographic Evaluation Of Lesion Sterilization And Tissue Repair Versus Zinc Oxide And Eugenol For Treatment of Necrotic Primary Molars
Brief Title: Lesion Sterilization And Tissue Repair Versus Zinc Oxide And Eugenol For Treatment of Necrotic Primary Molars
Acronym: LSTR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Ahmed Abdeltawab, principlal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSTR 3MIX-MP In Necrotic teeth
Record Dates: First submitted 2022-06-29; First posted 2022-07-08 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Necrotic Primary Molars
MeSH Terms: interventions — Wound Healing; Zinc Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 MIX (Experimental): Lesion sterilization and tissue repair; preparation of modified triple antibiotic paste tap: the chemotherapeutic agents used are metronidazole tablets 500 mg (flagyl®, sanofi, egypt), ciprofloxacin tablets 500 mg (ciproxcin®,. Epico, egypt,), and doxycycline capsules 100 mg (doxymycin™ dt, el-nile pharmaceuticals, egypt).
  Interventions: Procedure: Lesion sterilization and tissue repair
- Zinc oxide and Eugenol Pulpectomy (Active Comparator): zinc oxide and eugenol (prevestdent pro™, egypt).
  Interventions: Procedure: zinc oxide and eugenol pulpectomy

INTERVENTIONS:
Procedure: Lesion sterilization and tissue repair — Pulp therapy for necrotic primary molars
  Arms: 3 MIX
Procedure: zinc oxide and eugenol pulpectomy — Pulp therapy for necrotic primary molars
  Arms: Zinc oxide and Eugenol Pulpectomy

SUMMARY:
The aim of this study is to evaluate the clinical and radiographic success of Lesion Sterilization And Tissue Repair [ LSTR] antibiotic paste versus Zinc Oxide and Eugenol pulpectomy in the treatment of non-vital primary molars.

DETAILED DESCRIPTION:
Primary teeth with infected root canals are a common problem, particularly in patients where the infection has reached the peri radicular tissues .

Among the pastes used in the pulp therapy of primary teeth with pulp necrosis, zinc oxide and eugenol paste has been a reference in dentistry since 1930. Endodontic treatment using zinc oxide and eugenol paste has shown satisfactory clinical and radiographic results, requires mechanical chemical preparation before filling root canals.

The main difficulties of endodontic treatment of primary molars are related to the anatomical complexity of the root canals and the long time needed to carry out the treatment. The additional difficulty involved in diagnosing root resorption is a limiting condition for determining the actual working length and instrumentation.

Other pastes have been studied, such as those containing antibiotics in their composition, thus dispensing with root canal instrumentation (such as lesion sterilization and tissue repair using triple antibiotic paste in treatment of non-vital primary molars.

Lesion sterilization and tissue repair using triple antibiotic paste has relevant clinical and radiographic success rates in treatment of non-vital primary molars.

ELIGIBILITY:
Inclusion Criteria:

* Children:

  1. Aged between 5 years and 7 years.
  2. With deep caries involving pulp in primary molars.
* Teeth:

  1. Necrotic teeth with or without periapical or furcal lesions.
  2. Primary molars with minimal root resorption not more than 1/3 of root.

Exclusion Criteria:

* Children:

  1. Children with systemic disease
  2. Previous history of allergy to antibiotics used in the study.
  3. Children that will not attend follow up.
* Teeth:

  1. Caries in primary teeth exhibiting pre-shedding mobility.
  2. Non restorable teeth.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Post oper3tive pain | 1 month
  Measured by verbal question to patient/parents
Post operative pain | 3 months
  Measured by verbal question to patient/parents
Post operative pain | 6 months
  Measured by verbal question to patient/parents
Tenderness | 1 month
  Percussion test using back of a dental mirror
Tenderness | 3 months
  Percussion test using back of a dental mirror
Tenderness | 6 months
  Percussion test using back of a dental mirror
Swelling /sinus tract or fistula | 1 month
  Visual examination
Swelling /sinus tract or fistula | 3 months
  Visual examination
Swelling /sinus tract or fistula | 6 months
  Visual examination
Tooth mobility | 1 month
  Mobility test
Tooth mobility | 3 months
  Mobility test
Tooth mobility | 6 months
  Mobility test

SECONDARY OUTCOMES:
Internal /External root resorption | 6 months
  Radiographic examination
Furcation involvement /radiolucency | 6 months
  Radiographic examination

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen X, Liu X, Zhong J. Clinical and radiographic evaluation of pulpectomy in primary teeth: a 18-months clinical randomized controlled trial. Head Face Med. 2017 Oct 27;13(1):12. doi: 10.1186/s13005-017-0145-1. PMID 29073902
- [Background] Luengo-Fereira J, Ayala-Jimenez S, Carlos-Medrano LE, Toscano-Garcia I, Anaya-Alvarez M. Clinical and Radiographic Evaluation of Formocresol and Chloramphenicol, Tetracycline and Zinc Oxide-Eugenol Antibiotic Paste in Primary Teeth Pulpotomies: 24 month follow up. J Clin Pediatr Dent. 2019;43(1):16-21. doi: 10.17796/1053-4625-43.1.4. Epub 2018 Oct 5. PMID 30289365
- [Background] Moura J, Lima M, Nogueira N, Castro M, Lima C, Moura M, Moura L. LSTR Antibiotic Paste Versus Zinc Oxide and Eugenol Pulpectomy for the Treatment of Primary Molars with Pulp Necrosis: A Randomized Controlled Trial. Pediatr Dent. 2021 Nov 15;43(6):435-442. PMID 34937613
- [Background] Navit S, Jaiswal N, Khan SA, Malhotra S, Sharma A, Mukesh, Jabeen S, Agarwal G. Antimicrobial Efficacy of Contemporary Obturating Materials used in Primary Teeth- An In-vitro Study. J Clin Diagn Res. 2016 Sep;10(9):ZC09-ZC12. doi: 10.7860/JCDR/2016/21883.8426. Epub 2016 Sep 1. PMID 27790570
- [Background] Pramila R, Muthu MS, Deepa G, Farzan JM, Rodrigues SJ. Pulpectomies in primary mandibular molars: a comparison of outcomes using three root filling materials. Int Endod J. 2016 May;49(5):413-21. doi: 10.1111/iej.12478. Epub 2015 Jul 4. PMID 26059708
- [Background] Coll JA, Dhar V, Vargas K, Chen CY, Crystal YO, AlShamali S, Marghalani AA. Use of Non-Vital Pulp Therapies in Primary Teeth. Pediatr Dent. 2020 Sep 15;42(5):337-349. PMID 33087217
- [Background] Zacharczuk GA, Toscano MA, Lopez GE, Ortolani AM. Evaluation of 3Mix-MP and pulpectomies in non-vital primary molars. Acta Odontol Latinoam. 2019 Apr 1;32(1):22-28. PMID 31206571
- [Background] Smail-Faugeron V, Glenny AM, Courson F, Durieux P, Muller-Bolla M, Fron Chabouis H. Pulp treatment for extensive decay in primary teeth. Cochrane Database Syst Rev. 2018 May 31;5(5):CD003220. doi: 10.1002/14651858.CD003220.pub3. PMID 29852056